CLINICAL TRIAL: NCT01741701
Title: A Pilot Double-Blind, Parallel Group, Placebo Controlled Study of Oxaloacetate in Subjects With Treated Parkinson's Disease (PD)
Brief Title: A Pilot Study of Oxaloacetate in Subjects With Treated PD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Terra Biological LLC (Industry)
Responsible Party: Principal Investigator, Rajesh Pahwa, MD, Professor, Director PD and Movement Disorder Center, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13397
Record Dates: First submitted 2012-12-01; First posted 2012-12-05 (Estimated); Results first posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Oxaloacetic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxaloacetate (OAA) (Experimental): active capsule containing 100 mg OAA and 100 mg ascorbate, taken daily
  Interventions: Drug: Oxaloacetate (OAA)
- Placebo (Placebo Comparator): placebo capsules that contain only 100 mg ascorbate, taken daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxaloacetate (OAA)
  Other Names: benaGene™
  Arms: Oxaloacetate (OAA)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if Oxaloacetate (OAA) is a safe and effective treatment for Parkinson's disease. Each subject will be asked to make 3 study visits and complete two safety follow-up phone calls over a 4 month period.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent and follow instructions per the protocol
* Diagnosis of idiopathic PD within 7 years of diagnosis
* Taking stable doses of levodopa and would not predictably need adjustment in PD medications for 4 months
* Unified Parkinson's Disease Rating Scale (UPDRS) II + III at least 30 points at baseline

Exclusion Criteria:

* Previously taken Oxaloacetate
* Participation in other drug studies or use of other investigational products within 30 days prior to baseline
* In the Investigator's opinion, any unstable or clinically significant condition that would impair the subjects' ability to comply with study follow-up
* Other known or suspected cause of parkinsonism

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Pahwa, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxaloacetate (OAA): active capsule containing 100 mg OAA and 100 mg ascorbate, taken daily
  Oxaloacetate (OAA)
- Placebo: placebo capsules that contain only 100 mg ascorbate, taken daily
  Placebo
Period: Overall Study
Arm/Group | Oxaloacetate (OAA) | Placebo
Started | 18 | 15
Completed | 13 | 13
Not Completed | 5 | 2
Not completed — Adverse Event | 5 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxaloacetate (OAA) | Placebo | Total
Number analyzed (Participants) | 18 | 15 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (11.4) | 64.6 (9.4) | 63.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 15 | 14 | 29
Region of Enrollment [Number; unit: participants]
  United States | 18 | 15 | 33
PD Duration [Mean (Standard Deviation); unit: years] | 2.9 (1.5) | 3.1 (1.7) | 3.0 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Total Score
Description: The UPDRS has 3 subscales including Mentation (4 questions based on patient report with answers on a scale of 0-4, with a total of 16 points), Activities of Daily Living (13 questions based on patient report with answers on a scale of 0-4, with a total of 52 points) and Motor (27 questions based on clinician assessment on a scale of 0-4, with a total of 108 points). The total scores represents the sum of each of these sections for a total of 176 points with a higher score representing greater dysfunction.
Time Frame: 4 months
Population: Only subjects that completed the study were included in the efficacy analyses, those that withdrew were not included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxaloacetate (OAA) | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale
  UPDRS Total Score at Baseline | 41.1 (6.7) | 42.9 (10.8)
  UPDRS Total Score at 4 months | 34.9 (10.4) | 34.4 (12.4)
Statistical Analysis 1: Comparison: Oxaloacetate (OAA) vs Placebo; Test type: Superiority or Other; p = 0.50, t-test, 2 sided

2. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) ADL + Motor Score
Description: The UPDRS has 3 subscales including Mentation (4 questions based on patient report with answers on a scale of 0-4, with a total of 16 points), Activities of Daily Living (13 questions based on patient report with answers on a scale of 0-4, with a total of 52 points) and Motor (27 questions based on clinician assessment on a scale of 0-4, with a total of 108 points). This measure examined the ADL + Motor subscales which have a total of 160 points with a higher score representing greater dysfunction.
Time Frame: 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxaloacetate (OAA) | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale
  UPDRS ADL + Motor at Baseline | 39.4 (6.9) | 42.2 (10.7)
  UPDRS ADL + Motor at 4 months | 33.4 (10.2) | 33.9 (11.7)
Statistical Analysis 1: Comparison: Oxaloacetate (OAA) vs Placebo; Comparison of change between groups from baseline to 4 months; Test type: Superiority or Other; p = 0.51, t-test, 2 sided

3. Secondary Outcome: Parkinson's Disease Questionnaire - 39 (PDQ-39)
Description: The PDQ-39 is a measure of quality of life in Parkinson's disease patients. It has 39 questions each with a response from 0-4 for a total of 156 points. The total score is calculated as a percentage so the scores of the 39 items are added and divided by 156 and multiplied by 100. The higher the score the worse quality of life.
Time Frame: 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total possible score
Arm/Group | Oxaloacetate (OAA) | Placebo
Number analyzed (Participants) | 13 | 13
percentage of total possible score
  PDQ-39 Total Score at Baseline | 13.0 (8.9) | 10.1 (7.8)
  PDQ-39 total score at 4 months | 14.4 (11.2) | 11.3 (7.4)
Statistical Analysis 1: Comparison: Oxaloacetate (OAA) vs Placebo; Comparison between groups in the change from baseline to 4 months; Test type: Superiority or Other; p = 0.97, t-test, 2 sided

4. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: The MoCA is an assessment of cognitive function. The total possible score ranges from 0 to 30 points with a lower score representing greater cognitive impairment.
Time Frame: 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxaloacetate (OAA) | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale
  MoCA at Baseline | 27.4 (2.0) | 27.2 (2.4)
  MoCA at 4 months | 28.1 (1.6) | 27.6 (2.4)
Statistical Analysis 1: Comparison: Oxaloacetate (OAA) vs Placebo; Comparison between groups in the change from baseline to 4 months; Test type: Superiority or Other; p = .77, t-test, 2 sided

5. Secondary Outcome: Geriatric Depression Scale (GDS)
Description: The GDS is a measure of depression. The scale has 30 yes/no questions. Each question has a maximum score of 1 and a total possible score ranging from 0 to 30. The higher the score the greater the depression.
Time Frame: 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxaloacetate (OAA) | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale
  GDS at Baseline | 5.3 (4.4) | 3.3 (3.1)
  GDS at 4 months | 5.8 (5.4) | 3.8 (3.7)
Statistical Analysis 1: Comparison: Oxaloacetate (OAA) vs Placebo; Comparison between groups in change from baseline to 4 months; Test type: Superiority or Other; p = .90, t-test, 2 sided

6. Secondary Outcome: NonMotor Symptom Questionnaire (NMSQuest)
Description: The NMSQuest is a 30 item questionnaire with 30 yes/no questions. There is a total of 30 points with each "yes" score representing 1 point and therefore the higher the score the greater number of nonmotor symptoms present. The score can range from 0 to 30.
Time Frame: 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxaloacetate (OAA) | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale
  NMSQuest at Baseline | 7.1 (4.4) | 6.2 (4.4)
  NMSQuest at 4 months | 7.9 (6.3) | 6.9 (4.6)
Statistical Analysis 1: Comparison: Oxaloacetate (OAA) vs Placebo; Comparison between groups in change from baseline to 4 months; Test type: Superiority or Other; p = .95, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse effects for each subject were collected throughout the 4 month study period
Arm/Group | Oxaloacetate (OAA) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/15
Other Adverse Events (participants affected / at risk) | 11/18 | 4/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaloacetate (OAA) (N=18) | Placebo (N=15)
insomnia/stimulant (General disorders) | 3 (3) | 1 (1) — Subjects had difficulty sleeping and felt jittery - described as a stimulant effect by one
Worsening of Parkinson's disease (Nervous system disorders) | 7 (7) | 1 (1)
GI upset (Gastrointestinal disorders) | 4 (4) | 0 (0)
Fatigue (Nervous system disorders) | 2 (2) | 0 (0)
dizziness (General disorders) | 1 (1) | 0 (0)
Cognitive worsening (Psychiatric disorders) | 1 (1) | 1 (1)
Increased urination (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes